CLINICAL TRIAL: NCT06336187
Title: European Active Surveillance of Renal Cell Carcinoma Study (EASE RCC Study)
Acronym: EASE
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Alessandro Volpe, Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: UPO 2020 02
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Renal Cell Carcinoma
Keywords: active surveillance; small renal masses
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — prostate biopsy, blood sample, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RCC (renal cell carcinoma): Patients with small, incidentally detected, histologically confirmed renal cell carcinoma
  Interventions: Other: active surveillance; Genetic: molecular investigation

INTERVENTIONS:
Other: active surveillance — Follow-up visits will be scheduled 3 (optional) and 6 months after diagnosis, every 6 months up to 3 years and yearly thereafter.
Genetic: molecular investigation — Transcriptomic analysis of tissues

SUMMARY:
The goal of this observational, prospective, multi-national clinical study is to assess overall survival of patients who are diagnosed with incidental, histologically (biopsy) confirmed, <4 cm Renal Cell Carcinoma (RCC) and are managed conservatively with active surveillance.

The primary endpoint is overall survival. The Secondary endpoints are tumor growth rate, progression rate, cancer-specific survival, progression-free survival, identification of clinical and pathological variables and molecular and genetic markers that correlate with growth rate and progression.

The main question it aims to answer is: patients with RCC (less than 4 cm) diagnosis can be managed with active surveillance instead treated with invasive curative procedure? For all participants a percutaneous biopsy of the renal mass will be arranged in all cases to histologically confirm the diagnosis of RCC (unless a diagnostic biopsy has been acquired in the previous 6 months). As a minimum, two samples will be used for diagnostic purposes while remaining core(s) will be preserved for molecular studies.

Then, all patients will be under active surveillance, which is defined as the initial monitoring of tumor size by serial abdominal imaging (US, CT, or MRI) Follow-up visits will be scheduled 3 (optional) and 6 months after diagnosis, every 6 months up to 3 years and yearly thereafter. A follow-up visit will also be carried out at the time of progression when it occurs. Follow-up visits will include medical history and physical examination (optional), and assessment of concurrent medications, blood and urine collection and storage if participating in translational activities, cross-sectional abdominal and chest imaging exams.

Follow-up percutaneous biopsies of the renal tumor are not mandatory, but can be performed when considered clinically important.

DETAILED DESCRIPTION:
Rationale: Active surveillance can be considered a reasonable strategy for elderly patients with small renal tumors or patients with significant comorbidities who are not good surgical candidates. However, most available studies on active surveillance include small renal tumors that were not histologically confirmed as renal cell carcinoma (RCCs), including a proportion of benign tumors. Furthermore, follow-up protocol and indications to delayed intervention during active surveillance have not been generally standardized. There is a clear need of information on the growth rate and oncological outcomes of histologically confirmed RCCs by percutaneous biopsy at diagnosis and on the results of a standardized protocol of active surveillance of small RCCs.

Furthermore, if the measurement of tumor growth rate seems to be helpful for initial conservative management of patients with incidentally diagnosed small renal tumors, it is necessary to identify reliable genetic or molecular serum, urine or tissue markers that can differentiate small renal tumors with different inherent aggressiveness and metastatic potential at diagnosis, thereby enabling the urologist to choose the most suitable conservative or active, individualized management approach for each patient.

This is a prospective, multi-national clinical study conducted in European countries by hospital based urologists. A total of 400 patients with small, incidentally detected, histologically confirmed RCCs will be included and data related to the oncological outcomes of an active surveillance approach will be collected.

After ethics committee approval, according to local requirements, and written patient informed consent has been obtained, patient enrolment can be started.

Primary endpoint is overall survival. Secondary endpoints are tumor growth rate, progression rate, cancer-specific survival, progression-free survival, identification of clinical and pathological variables and molecular and genetic markers that correlate with growth rate and progression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age ≥ 18 years
* Incidental diagnosis at imaging (ultrasonography, CT, MRI) of a solid renal mass < 4 cm in maximum diameter.
* Histologically confirmed RCC by percutaneous needle biopsy at diagnosis. All RCC subtypes are eligible for the study.
* Patients unfit for active treatment due to advanced age, or co-morbidity, or choosing to avoid active treatment.
* Signed Informed consent.
* Preparedness to comply with percutaneous tumor biopsy and a close follow-up protocol

Exclusion Criteria:

* Renal tumors with a non-RCC histology (sarcomas, lymphomas, etc.).
* Presence of metastatic disease at diagnosis
* Tumor related symptoms at presentation.
* Patients with known genetic diseases associated with RCC (Von Hippel-Lindau, Birt-Hogg-Dubé, Hereditary Leiomyomatosis and Renal Cell Cancer, etc.).
* Patients unsuitable for biopsy due to need for concomitant anticoagulation or anti-platelet drug use which cannot be transiently discontinued.
* Patients unsuitable for biopsy due to tumor location or small tumor size.
* Patients with concurrent systemic treatment for another cancer.
* Patients with estimated life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multi-national clinical study conducted in European countries by hospital based urologists. Patients with small, incidentally detected, histologically confirmed renal cell carcinoma will be included and data related to the oncological outcomes of an active surveillance approach will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | more than 3 years
  Overall survival

SECONDARY OUTCOMES:
Disease progression | more than 3 years
  tumor growth rate, progression rate, cancer-specific survival, progression-free survival
Molecular pattern | more than 3 years
  identification of molecular and genetic markers that correlate with growth rate and progression

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided